CLINICAL TRIAL: NCT01337193
Title: Effect of Rehabilitative Ultrasound Imaging Biofeedback on Urinary Incontinence, Pelvic Floor Muscle Contractions and Quality of Life in Women With Stress Urinary Incontinence
Brief Title: Effect of Exercise and Biofeedback on Symptoms of Incontinence in Women With Stress Urinary Incontinence
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal investigator has decided not to continue her PhD studies.
Sponsor: Texas Woman's University (Other)
Responsible Party: Principal Investigator, Elaine Trudelle-Jackson, PhD Advisor, Texas Woman's University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SUI 16333
Record Dates: First submitted 2011-04-01; First posted 2011-04-18 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Stress Urinary Incontinence
Keywords: stress urinary incontinence; exercise; pelvic floor muscles; biofeedback; rehabilitative ultrasound imaging
MeSH Terms: conditions — Urinary Incontinence, Stress; Motor Activity | interventions — Biofeedback, Psychology

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pelvic floor muscle exercises (Active Comparator): Three pelvic floor muscle exercises will be performed with verbal cueing from the instructor.
  Interventions: Other: Pelvic floor muscle exercises
- Pelvic floor exercises with biofeedback (Experimental): Pelvic floor exercises will be performed with biobeedback cueing.
  Interventions: Other: Pelvic floor exercises with biofeedback

INTERVENTIONS:
Other: Pelvic floor exercises with biofeedback — Exercises will be performed with assistance of biofeedback cueing
  Arms: Pelvic floor exercises with biofeedback
Other: Pelvic floor muscle exercises — Exercises will b performed with verbal cueing of investigator.
  Arms: Pelvic floor muscle exercises

SUMMARY:
The overall purpose of this research is to determine the effect of ultrasound imaging biofeedback on urine leakage, pelvic floor muscle contractions, and quality of life in women with stress urinary incontinence. This study will include women 20 years or older with stress urinary incontinence.

The study will involve 2 groups: pelvic floor muscle (PFM) exercises with biofeedback using transabdominal Rehabilitative ultrasound imaging (RUSI) (Group A) and PFM exercises alone (Group B). The participants will perform 16 exercise sessions over a period of 8 weeks. Group A will perform 3 pelvic floor exercises using the transabdominal RUSI to provide biofeedback. Group B will perform the same 3 pelvic floor exercises without biofeedback.

All participants involved in the study will complete a general medical information questionnaire. In addition, all participants will have their PFM contraction assessed using an ultrasound machine placed over the lower abdomen, quality of life assessed with a written questionnaire, and given a 7-day bladder diary to complete prior to, at 4-weeks, and at completion of the study.

DETAILED DESCRIPTION:
This study has been terminated.

ELIGIBILITY:
Inclusion Criteria:

1. women will need to be 20 years or older
2. diagnosed with stress urinary incontinence (SUI).

Exclusion Criteria:

women with:

1. urge or mixed incontinence
2. pelvic organ prolapse
3. previous surgical treatment for incontinence
4. current treatment for SUI (including medications)
5. current pregnancy
6. six months or less postpartum
7. body mass index of ≥ 30
8. recurrent vulvovaginitis
9. current/recurrent urinary tract infections (UTI)
10. non-English speaking.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change in the ability to contract the pelvic floor muscles from baseline to the midpoint and completion of the study | baseline, 4 weeks, and 8 weeks
  Pelvic floor muscle lift and length of pelvic floor muscle contraction will be measured using transabdominal ultrasound imaging. Ability to maintain continence during a cough will be measured by asking the participant to stand, contract the pelvic floor muscles, and cough. The participant will state whether or not they leaked urine.

SECONDARY OUTCOMES:
Change in the number of incontinent episodes per week from baseline to the midpoint and conclusion of the study | Baseline, 4 weeks, and 8 weeks
  Incidence of incontinent episodes will be measured using a 7-day bladder diary
Change in quality of life from the baseline to the midpoint and completion of the study | Baseline, 4 weeks, and 8 weeks
  Quality of life will be measured using the I-QOL questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Trudell-Jackson, PT, PhD, Study Chair — Texas Woman's University
Locations (1):
- Texas Woman's University, Dallas, Texas, United States